CLINICAL TRIAL: NCT06885957
Title: A Registry Study on Monoclonal Antibody-Based Therapies for Aquaporin-4 Antibody-Positive Neuromyelitis Optica Spectrum Disorders
Brief Title: Monoclonal Antibody-Based Therapies for AQP4-Positive NMOSD
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Daishi Tian, Professor, Tongji Hospital
Other Study IDs: MabInNMOSD
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: NMO Spectrum Disorder
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Inebilizumab treatment: AQP4-IgG positive NMOSD Patient who received Inebilizumab
  Interventions: Drug: Mab Therapy
- Satralizumab treatment: AQP4-IgG positive NMOSD Patient who received Satralizumab
  Interventions: Drug: Mab Therapy
- Eculizumab treatment: AQP4-IgG positive NMOSD Patient who received Eculizumab
  Interventions: Drug: Mab Therapy
- Ofatumumab treatment: AQP4-IgG positive NMOSD Patient who received Ofatumumab
  Interventions: Drug: Mab Therapy
- Rituximab treatment: AQP4-IgG positive NMOSD Patient who received Rituximab
  Interventions: Drug: Mab Therapy
- Conventional immunosuppressive agents treatment: AQP4-IgG positive NMOSD Patient who received Conventional immunosuppressive agents

INTERVENTIONS:
Drug: Mab Therapy — Whether receive mab therapy or not.
  Groups: Eculizumab treatment; Inebilizumab treatment; Ofatumumab treatment; Rituximab treatment; Satralizumab treatment

SUMMARY:
The primary objective of this registry study is to evaluate the therapeutic efficacy and safety profiles of distinct monoclonal antibody-based therapies for aquaporin-4 immunoglobulin G-seropositive neuromyelitis optica spectrum disorders within the Chinese population under real-world clinical conditions. Secondary objectives include quantitative assessment of longitudinal neuroimaging biomarker variations and immunological profile alterations in longitudinal biological specimens pre- and post-therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must demonstrate capacity to comprehend the study's objectives and associated risks, provide written informed consent, and authorize utilization of confidential health information in compliance with national and regional data protection regulations.
* Enrollment is permitted regardless of biological sex, with age ≥18 and ≤65 years (inclusive) at the time of informed consent provision.
* All females of childbearing potential and biologically male participants must employ contraceptive measures meeting clinical trial standards throughout the study duration and for at least 30 days following the final administration of investigational therapy. Additionally, participants must abstain from gamete donation during the study period and for ≥30 days post-treatment cessation.
* Confirmed diagnosis of aquaporin-4 immunoglobulin G (AQP4-IgG)-seropositive neuromyelitis optica spectrum disorders (NMOSD) per the 2015 International Consensus Diagnostic Criteria, with serological or cerebrospinal fluid verification of AQP4-IgG positivity for inclusion in the AQP4-NMOSD cohort. Participants must have provided documented consent for therapeutic intervention with one monoclonal antibody-based biologics.
* Neurological examination demonstrating clinical stability within 30 days preceding baseline (Visit 1).

Exclusion Criteria:

* Medical History and Current Health Status

  1. Clinically significant medical history of cardiac, endocrine, hematologic, hepatic, immune, infectious, metabolic, renal, pulmonary, neurological, dermatologic, psychiatric, or other major systemic conditions that, in the investigator's judgment, would preclude safe trial participation.
  2. Prior cerebrovascular events resulting in a baseline modified Rankin Scale (mRS) score >3.
  3. Hypersensitivity to the investigational therapeutic agent(s) or their excipients.
* Infection Risk

  1. Documented history or positive screening test for human immunodeficiency virus (HIV).
  2. Active hepatitis C virus (HCV) infection, defined as detectable HCV RNA with concomitant anti-HCV antibody positivity. Subjects with anti-HCV antibody positivity and undetectable HCV RNA remain eligible.
  3. Active hepatitis B virus (HBV) infection, defined as hepatitis B surface antigen (HBsAg) positivity and/or total hepatitis B core antibody (anti-HBc) positivity. Subjects with prior natural infection (HBsAg-negative, anti-HBc-positive, and anti-HBs-positive) or vaccination-induced immunity (HBsAg-negative, anti-HBc-negative, and anti-HBs-positive) are eligible.
  4. Chronic, recurrent, or severe infections (e.g., pneumonitis, sepsis) within 90 days prior to baseline (Visit 1).
  5. History of active tuberculosis (TB) or latent TB infection, defined by positive interferon-gamma release assay (IGRA) results or two consecutive tuberculin skin tests.
  6. Active bacterial, fungal, or viral infections (including upper respiratory tract infections) within 28 days prior to baseline. Subjects with localized fungal infections (e.g., candidiasis, dermatophytosis) may undergo re-screening post-treatment.
  7. Contraindications to rescue therapies, including rituximab, intravenous immunoglobulin (IVIG), high-dose corticosteroids, or cyclophosphamide.
  8. Prior exposure to total lymphoid irradiation, cladribine, T-cell or T-cell receptor vaccination, total body irradiation, or hematopoietic stem cell transplantation at any time.
* Additional Exclusion Criteria

  1. Clinically significant suicidal ideation or behavior within the past 12 months, as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS).
  2. Unwillingness or inability to comply with protocol-mandated procedures.
  3. Severe auditory/visual impairment, language barriers, claustrophobia, or other conditions precluding neuropsychological assessments or MRI completion.
  4. Any other condition deemed by the investigator or sponsor to compromise subject eligibility or study integrity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Confirmed diagnosis of aquaporin-4 immunoglobulin G (AQP4-IgG)-seropositive neuromyelitis optica spectrum disorders (NMOSD) per the 2015 International Consensus Diagnostic Criteria, with serological or cerebrospinal fluid verification of AQP4-IgG positivity for inclusion in the AQP4-NMOSD cohort.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to first relapse | Up to 96 weeks
Median time to relapse | Up to 96 weeks
Annualized relapse rate | Up to 96 weeks
EDSS score | Up to 96 weeks

SECONDARY OUTCOMES:
Incidence of radiologically identified new gadolinium-enhancing lesions and/or new or enlarging T2-weighted lesions | Up to 96 weeks
AQP4-IgG titer in serum and cerebral spinal fluid | Up to 96 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No